CLINICAL TRIAL: NCT03148912
Title: Optimizing the Diagnosis of Heparin Induced Thrombocytopenia Using Quantified Anti-Platelet Factor 4 Immunological Testing: A Pilot Multicentre Cohort Study
Brief Title: Optimizing the Diagnosis of Heparin Induced Thrombocytopenia
Acronym: HIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRIS6428
Record Dates: First submitted 2017-04-10; First posted 2017-05-11 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Heparin-induced Thrombocytopenia (HIT)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- diagnostic algorithm (Experimental): Optimizing the interpretation of the more readily available anti-PF4 assay would reduce the reliance on functional testing/ confirmatory testing (Serotonin Release Assay, SRA) and the number of patients exposed to unnecessary changes in anticoagulation therapy while awaiting the timely functional test results
  Interventions: Diagnostic Test: Diagnostic algorithm

INTERVENTIONS:
Diagnostic Test: Diagnostic algorithm — The treating physician will complete an enrollment assessment including the 4T score pretest probability assessment14. All patients will have laboratory testing for HIT anti-PF4 as well as SRA testing. Results of the anti-PF4 assay (OD value) will be available to the treating physician who will be instructed to follow the study diagnostic algorithm

SUMMARY:
Multicentre (Ottawa and Halifax) prospective cohort study using a diagnostic approach in patients clinically suspected to have HIT that combines pretest probability assessment with quantitative interpretation of anti-PF4 assay.

DETAILED DESCRIPTION:
The proposed is a prospective cohort study exploring a novel diagnostic approach to Heparin Induced Thrombocytopenia (HIT) using a combination of pretest probability assessment and quantitative interpretation of the anti-platelet factor 4 Immunological assay (anti-PF4). Patient with a clinical suspicion of HIT will follow the study diagnostic algorithm (Figure 1). The study algorithm will be considered a safe approach to move forward into a larger RCT if the upper limit of the 95% confidence interval for 'false negative management failures' is ≤ 4% based on a Serotonin Release Assay (SRA) gold standard. The main objective of the pilot study is to inform feasibility and recruitment barriers for a larger randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

* Patient with clinical suspicion of HIT by treating physician

Exclusion Criteria:

1. Less than 18 years of age;
2. Prior diagnosis of HIT ever;
3. Patient enrolled within preceding 100 days;
4. Functional/ confirmatory platelet activation results available at the time of enrollment;
5. Requiring cardio-pulmonary bypass or percutaneous cardiac angioplasty or any other cardiac or vascular surgery/procedure requiring intra-operative/procedural heparin administration planned within 30 days;
6. Unable to complete study follow up;
7. Unable to obtain consent (or proxy consent from substitute decision maker where applicable);
8. Life expectancy less than 30 days;
9. Greater than 72 hours from clinical suspicion of HIT and/or request for HIT anti-PF4 ELISA testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-11-23 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Recruitment | 2 years
  The pilot will be considered feasible if recruitment of at least 7.5 patients per month (total between the two sites) is achieved.
False negative management failures | 2 years
  The rate of false negative 'management failures' where the study protocol concludes HIT unlikely but SRA (reference standard laboratory test) is positive for HIT (≥50% Serotonin release).

SECONDARY OUTCOMES:
Major arterial and venous thromboembolism events | 24 hours of baseline and 24 of study enrolment
  Events will be ascertained from the date of study consent. However, venous or arterial thrombotic events detected on investigations ordered within 24 hours of study entry will be captured as baseline events and will be counted separately from thrombotic events which occur after the initial 24 hours of study enrolment.
Proximal deep vein thrombosis | 2 years
  Testing performed because of symptoms in a patient with (new) non-compressibility of the common femoral vein, popliteal vein or calf trifurcation vein of the leg on ultrasound; or new non-compressibility or visualization of thrombus in the jugular vein, subclavian vein or axillary vein on ultrasound; or an intraluminal defect seen in one more than one view in proximal leg or arm veins on venography will be diagnostic for deep vein thrombosis.
Pulmonary embolism | 2 years
  Testing performed because of symptoms in a patient with a high probability lung scan (i.e. at least one segmental perfusion mismatch) or CT pulmonary angiography (i.e. intraluminal filling defect in the main, lobar or segmental pulmonary arteries) will be diagnostic for pulmonary embolism.
Stroke | 2 years
  New infarction or hemorrhagic event confirmed on CT or MRI.
Myocardial infarction | 2 years
  Detection of rise and/or fall of cardiac biomarkers (preferably troponin) with at least one value above the 99th percentile of the upper reference limit together with evidence of myocardial ischemia with at least one of the following: Symptoms of ischemia for ≥ 20 minutes ECG changes indicative of new ischemia: new ST-T changes ≥0.1 mV or new left bundle branch block Development of pathological Q waves in the ECG; Imaging evidence of new loss of viable myocardium or new regional wall motion abnormality.
Systemic arterial embolism | 2 years
  Acute vascular occlusion confirmed on ultrasound or angiography Adrenal hemorrhagic infarction (indicating adrenal vein thrombosis) - radiologic diagnosis on ultrasound or CT.
Death | 30 days of follow up
  Due to major arterial or venous thromboembolism within 30days of follow up and major and minor bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Duffett, MSc, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Linkins LA, Dans AL, Moores LK, Bona R, Davidson BL, Schulman S, Crowther M. Treatment and prevention of heparin-induced thrombocytopenia: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e495S-e530S. doi: 10.1378/chest.11-2303. PMID 22315270
- [Background] Raschke RA, Curry SC, Warkentin TE, Gerkin RD. Improving clinical interpretation of the anti-platelet factor 4/heparin enzyme-linked immunosorbent assay for the diagnosis of heparin-induced thrombocytopenia through the use of receiver operating characteristic analysis, stratum-specific likelihood ratios, and Bayes theorem. Chest. 2013 Oct;144(4):1269-1275. doi: 10.1378/chest.12-2712. PMID 23703622
- [Background] Greinacher A, Ittermann T, Bagemuhl J, Althaus K, Furll B, Selleng S, Lubenow N, Schellong S, Sheppard JI, Warkentin TE. Heparin-induced thrombocytopenia: towards standardization of platelet factor 4/heparin antigen tests. J Thromb Haemost. 2010 Sep;8(9):2025-31. doi: 10.1111/j.1538-7836.2010.03974.x. PMID 20626620
- [Background] Warkentin TE. How I diagnose and manage HIT. Hematology Am Soc Hematol Educ Program. 2011;2011:143-9. doi: 10.1182/asheducation-2011.1.143. PMID 22160026
- [Background] Zwicker JI, Uhl L, Huang WY, Shaz BH, Bauer KA. Thrombosis and ELISA optical density values in hospitalized patients with heparin-induced thrombocytopenia. J Thromb Haemost. 2004 Dec;2(12):2133-7. doi: 10.1111/j.1538-7836.2004.01039.x. PMID 15613017
- [Background] Lo GK, Sigouin CS, Warkentin TE. What is the potential for overdiagnosis of heparin-induced thrombocytopenia? Am J Hematol. 2007 Dec;82(12):1037-43. doi: 10.1002/ajh.21032. PMID 17722079
- [Background] Warkentin TE. HIT paradigms and paradoxes. J Thromb Haemost. 2011 Jul;9 Suppl 1:105-17. doi: 10.1111/j.1538-7836.2011.04322.x. PMID 21781246
- [Background] Warkentin TE, Greinacher A, Gruel Y, Aster RH, Chong BH; scientific and standardization committee of the international society on thrombosis and haemostasis. Laboratory testing for heparin-induced thrombocytopenia: a conceptual framework and implications for diagnosis. J Thromb Haemost. 2011 Dec;9(12):2498-500. doi: 10.1111/j.1538-7836.2011.04536.x. No abstract available. PMID 22947414
- [Background] Warkentin TE, Sheppard JI, Moore JC, Sigouin CS, Kelton JG. Quantitative interpretation of optical density measurements using PF4-dependent enzyme-immunoassays. J Thromb Haemost. 2008 Aug;6(8):1304-12. doi: 10.1111/j.1538-7836.2008.03025.x. Epub 2008 May 17. PMID 18489711
- [Background] Linkins LA, Bates SM, Lee AY, Heddle NM, Wang G, Warkentin TE. Combination of 4Ts score and PF4/H-PaGIA for diagnosis and management of heparin-induced thrombocytopenia: prospective cohort study. Blood. 2015 Jul 30;126(5):597-603. doi: 10.1182/blood-2014-12-618165. Epub 2015 Apr 29. PMID 25926600
- [Background] Lo GK, Juhl D, Warkentin TE, Sigouin CS, Eichler P, Greinacher A. Evaluation of pretest clinical score (4 T's) for the diagnosis of heparin-induced thrombocytopenia in two clinical settings. J Thromb Haemost. 2006 Apr;4(4):759-65. doi: 10.1111/j.1538-7836.2006.01787.x. PMID 16634744
- [Background] Thygesen K, Alpert JS, White HD; Joint ESC/ACCF/AHA/WHF Task Force for the Redefinition of Myocardial Infarction. Universal definition of myocardial infarction. J Am Coll Cardiol. 2007 Nov 27;50(22):2173-95. doi: 10.1016/j.jacc.2007.09.011. No abstract available. PMID 18036459
- [Background] Schulman S, Kearon C; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in non-surgical patients. J Thromb Haemost. 2005 Apr;3(4):692-4. doi: 10.1111/j.1538-7836.2005.01204.x. PMID 15842354